CLINICAL TRIAL: NCT03410953
Title: Vaccination Adjuved Against Hepatitis B in SNS Workers Typed as no Responders to Conventional Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other); Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IBS-VACANTIB-1701; 2016-004991-23 (EudraCT Number); GRS1360/A/16 (Other Grant/Funding Number: G.R.Salud de Castilla y León, Junta CyL); 17/1311 (Other: IBSAL (INSTITUTO DE INVESTIGACION BIOMEDICA DE SALAMANCA))
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis B; Hepatitis; Hepatitis, Viral, Human; Hepatitis B Immunization
MeSH Terms: conditions — Hepatitis B; Hepatitis; Hepatitis, Viral, Human | interventions — DNA, Ribosomal; Vaccines

STUDY DESIGN:
Intervention Model Description: non-responders to conventional treatment of hepatitis B vaccination and consent to participate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fendrix (Experimental): The primary immunisation consists of 4 separate 0.5 ml doses of FENDRIX administered at the following schedule:
  1 month, 2 months and 6 months from the date of the first dose. Once initiated, the primary course of vaccination at 0, 1, 2 and 6 months should be completed with Fendrix, and not with other commercially available HBV vaccine
  Interventions: Biological: Fendrix suspension for injection Hepatitis B (rDNA) vaccine (adjuvanted, adsorbed).

INTERVENTIONS:
Biological: Fendrix suspension for injection Hepatitis B (rDNA) vaccine (adjuvanted, adsorbed). — The primary immunisation consists of 4 separate 0.5 ml doses administered at the following schedule:
  1 month, 2 months and 6 months from the date of the first dose. Once initiated, the primary course of vaccination at 0, 1, 2 and 6 months should be completed with Fendrix, and not with other commercially available HBV vaccine

SUMMARY:
Health workers with biological risk in their tasks, who have been vaccinated as non-responders to conventional vaccination against Hepatitis B. To provide Health workers-staff with an additional protection tool against hepatitis B infection. To evaluate the efficacy of the adjuvanted vaccine in healthy nonresponders to conventional hepatitis B vaccine.

DETAILED DESCRIPTION:
An interventional, phase 4, single group assignment, without masking (open label), preventive clinical trial was carried out in health workers with biological risk in their tasks, who have been filed as non-responders to conventional vaccination against Hepatitis B.

Methods: 67 health workers with biological risk in their tasks, who have been filed as non-responders to conventional vaccination against Hepatitis B, were enrolled in the Clinical Trial. All participants were from 18 years up to 64 years old. The criteria defining them as non-responders to the conventional hepatitis B vaccine is anti HBsAb titers < 10 mUI/ml following the application of six doses of conventional vaccine at 20 lg doses (two complete guidelines). The objective of this study was to provide Health workersstaff with an additional protection tool against hepatitis B infection, and to evaluate the efficacy of the adjuvanted vaccine in healthy non-responders to conventional hepatitis B vaccine.

ELIGIBILITY:
Inclusion Criteria:

* NHS workers -including university students doing their internships in health centres dependent on the National Health System (inclusion of students is regulated and limited by specific instructions on labour prevention in each autonomous community).
* Criteria defining them as NO responders to the conventional hepatitis B vaccine: anti HBsAb titers <10 mIU / ml following the application of six doses of conventional vaccine at 20 μg doses (two complete guidelines).

Exclusion Criteria:

* Known allergy to the active substance or any of the other ingredients of the medicinal product (included in section 6 of the product data sheet).
* Subjects that have ever had an allergic reaction to any vaccine against hepatitis B.
* Subjects have a serious infection with fever.
* Subjects for whom informed consent is not obtained.
* Subjects that have not revoked the consent initially signed.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose L. Bravo-Grande, MD PhD, Principal Investigator — IBSAL-Instituto de Investigación Biomédica de Salamanca
Locations (11):
- Spain (11):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Asistencial Universitario de Palencia, Palencia
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Complejo Asistencial de Zamora, Zamora

REFERENCES:
- [Derived] Bravo-Grande JL, Asuncion Blanco-Gonzalez M, de la Torre-Robles JM, Asmat-Inostrosa MP, Fernandez-Escribano M, Villalobos IM, Covadonga Caso-Pita M, Hervella-Ordonez M, Canibano Cimas LM, de la Fuente-Martin JM, Luisa Rodriguez de la Pinta M, Olivas JRB, Munoz-Ruiperez C, Alonso Lopez MA, Del Campo MT, Antonieta Ramirez Perez M, Sanchez-Arcilla I, Marzola-Payares M, Rescalvo-Santiago F, Paula-Ortiz M, Sanchez-Santos JM, Lopez-Perez R. Vaccination adjuvated against hepatitis B in Spanish National Healthcare System (SNS) workers typed as non-responders to conventional vaccines. Vaccine. 2021 Jan 15;39(3):554-563. doi: 10.1016/j.vaccine.2020.12.006. Epub 2020 Dec 15. PMID 33334613

RESULTS

PARTICIPANT FLOW:
Groups:
- Fendrix: The primary immunisation consists of 4 separate 0.5 ml doses of FENDRIX administered at the following schedule:
  1 month, 2 months and 6 months from the date of the first dose. Once initiated, the primary course of vaccination at 0, 1, 2 and 6 months should be completed with Fendrix, and not with other commercially available HBV vaccine
  Fendrix suspension for injection Hepatitis B (rDNA) vaccine (adjuvanted, adsorbed).: The primary immunisation consists of 4 separate 0.5 ml doses administered at the following schedule:
  1 month, 2 months and 6 months from the date of the first dose. Once initiated, the primary course of vaccination at 0, 1, 2 and 6 months should be completed with Fendrix, and not with other commercially available HBV vaccine
Period: Overall Study
Arm/Group | Fendrix
Started | 67 (First patient recruited)
Completed | 67 (67 participants were enrolled in the Clinical Trial and included the analyses)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects had to work in the SNS -including university students undertaking work placements in SNS health centres (subject to and limited by the specific regulations on health and safety in each autonomous region)- and be of working age.
Arm/Group | Fendrix
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 67
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.46 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 67
Region of Enrollment [Number; unit: participants]
  Spain | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Protective Levels of Antibodies After Treatment
Description: Measurement of antibody antiHBs: before the first dose and a month after the administration of each dose.
Time Frame: Between 40 and 60 days after the last dose given
Measure: Count of Participants; unit: Participants
Arm/Group | Fendrix
Number analyzed (Participants) | 67
Participants
  Positive | 63
  Negative | 4

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: AE 32 SAE 0 Total 32
Arm/Group | Fendrix
All-Cause Mortality (participants affected / at risk) | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67
Other Adverse Events (participants affected / at risk) | 29/67
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fendrix (N=67)
Puncture Zone Pain (Skin and subcutaneous tissue disorders) | 19
Discomfort (General disorders) | 4
Fatigue (General disorders) | 3
Diarrhea (General disorders) | 2
Paresthesia in the puncture area (General disorders) | 2
Cramp (General disorders) | 1
Diverticulitis (General disorders) | 1

LIMITATIONS AND CAVEATS:
Number of possible participants from all hospitals were small. This resulted in the need to extend recruitment to additional centres in order to obtain an optimal study sample.

We also encountered a lack of information concerning staff who do not respond to vaccination.

We also encountered some isolated difficulties as regards organizing all trial visits and their dates for various reasons, including vacations and sick leave. It was resolved through study coordination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT03410953/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT03410953/ICF_001.pdf